CLINICAL TRIAL: NCT00732368
Title: A Long-term Study of Mometasone Furoate in Patients With Perennial Allergic Rhinitis
Brief Title: A Long-term Study of Mometasone Furoate in Patients With Perennial Allergic Rhinitis (Study P04459)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04459
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mometasone Nasal Spray (Experimental): Open-label. Two sprays per nostril once daily (200 mcg/day). After 4 weeks, dose can be decreased to one spray per nostril daily or increased to 4 sprays per nostril daily.
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: Mometasone furoate — Two sprays mometasone nasal spray per nostril once daily (200 mcg/day). After 4 weeks, dose can be decreased to one spray per nostril daily or increased to 4 sprays per nostril daily.
  Other Names: SCH 032088; Nasonex

SUMMARY:
This study examined the safety and effectiveness of long-term administration of mometasone nasal spray in patients with perennial allergic rhinitis. Patients received mometasone for 12 weeks plus an additional 12 weeks if patient agreed to continue. Dose of mometasone could be decreased or increased during the study based on patient's response.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe perennial allergic rhinitis, >16 years of age

Exclusion Criteria:

* Patients with coexisting tuberculous disease or lower respiratory tract infection and patients who have acute upper respiratory tract infection, acute pharyngolaryngitis, or acute tonsillitis judged by the investigator to require treatment
* Patients with coexisting infections or systemic mycosis for which there are no effective treatment
* Patients with coexisting mycosis in the nasal and paranasal cavities
* Patients who are judged to require prohibited concomitant drugs during the clinical study
* Patients who have experienced recent nasal septum ulcers, nasal surgery, or nasal trauma, which have not yet healed
* Patients with a history of hypersensitivity to steroids or mometasone furoate
* Patients who are pregnant or nursing or who may be pregnant and patients or whose partner desires to become pregnant during the study period
* Patients with severe hepatic disorder, renal disorder, cardiac disease, diabetes mellitus, hypertension, or hematological disease or other serious coexisting diseases and whose general condition is poor as judged by the investigators.
* Patients allergic to pollen and the pollen release season occurs in the 7 days before the start of treatment
* Patients diagnosed with vasomotor rhinitis or eosinophilic rhinitis
* Patients with nasal conditions which may interfere with efficacy evaluation of the study drug
* Patients who develop a disease which may affect nasal symptoms in the 7 days before the start of treatment
* Patients who are participating or have participated in a clinical trial of an investigational drug within 120 days before the day of obtaining informed consent
* Patients for whom the period of discontinuation of previous treatment before the start of study drug administration indicated Table 2 is not adequate or who cannot avoid the use of these drugs
* Patients undergoing specific desensitization therapy or nonspecific allassotherapy (Histaglobin, vaccine therapy, etc.) or who had discontinued such therapy within 90 days prior to obtaining informed consent. (However, patients need not be excluded if therapy has been ongoing for at least 180 days before obtaining informed consent and maintenance therapy is now being conducted.)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2006-01-01 (Actual); Study Completion 2006-01-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in 4 nasal symptom score. | All visits starting 2 weeks prior to treatment until 5 to 9 days after last administration of treatment

SECONDARY OUTCOMES:
Individual nasal symptom scores (sneezing, attack, rhinorrhea, nasal congestion, and nasal itching) | All visits starting 2 weeks prior to treatment until 5 to 9 days after last administration of treatment
Overall improvement (combination of nasal symptoms and rhinoscopic nasal findings) | All visits during which patient is receiving drug (includes the 12 week drug administration period plus the 12 week additional drug administration period)
Adverse events | Throughout the study once initial treatment has started and until 5 to 9 days after last administration of treatment.
Laboratory tests | At baseline, and 4, 12, and 24 weeks after treatment

REFERENCES:
- [Result] T. Ishikawa et. al; Practica otologica. Suppl. 122 Page1-17(2008.11) -Japanese language journal